CLINICAL TRIAL: NCT03979911
Title: Evaluation of Double HER2 Blocking by Pertuzumab-Trastuzumab and Taxane in the Standard Treatment of Metastatic Breast Cancer
Brief Title: Evaluation of Pertuzumab-Trastuzumab and Taxane in the Standard Treatment of Metastatic Breast Cancer
Acronym: EPTTCSM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: EPTTCSM (239BRC18.0129)
Record Dates: First submitted 2019-04-17; First posted 2019-06-07 (Actual); Last update posted 2019-06-07 (Actual); Status verified 2018-11

CONDITIONS: Breast Neoplasms; HER-2 Gene Amplification
Keywords: Pertuzumab; Breast Neoplasms/pathology; Real life; Trastuzumab; Receptor, ErbB-2/antagonists & inhibitors*; Breast Neoplasms/drug therapy*; Multicenter Study; Taxoids; Antibodies, Monoclonal, Humanized
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective study evaluated the efficacy and the safety of use of this treatment combined with a taxane for the treatment of HER2-positive metastatic breast cancer and compared the clinical and demographic characteristics of real life patients to the patients of CLEOPATRA.

DETAILED DESCRIPTION:
In 2013 the European Medicines Agency authorized the use of a new antibody named Pertuzumab in combination with Trastuzumab in first-line setting for patients with HER2-positive metastatic breast cancer. The efficacy and the safety were demonstrated in the CLEOPATRA study. This study had inclusion and exclusion criteria that might not be representative of a real life population of women with metastatic breast cancer. Few study tried to evaluate this treatment in real life settings but with discordant results. This retrospective study evaluated the efficacy and the safety of use of this treatment combined with a taxane for the treatment of HER2-positive metastatic breast cancer and compared the clinical and demographic characteristics of real life patients to the patients of CLEOPATRA.

ELIGIBILITY:
Inclusion Criteria:

* metastatic breast cancer
* HER2 positive
* Received pertuzumab in combination with trastuzumab and taxane chemotherapy

Exclusion Criteria:

* no HER2-positive breast cancer
* no association with taxane chemotherapy
* no metastatic breast cancer
* refusal to consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with metastatic breast cancer HER2 positive who received pertuzumab in combination with trastuzumab and taxane chemotherapy
Sampling Method: Non-Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-07-22 (Estimated); Study Completion 2019-07-22 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | through study completion, an average of 1 year
  time between inclusion and progression of the disease
overall survival | through study completion, an average of 1 year
  time between inclusion and death

SECONDARY OUTCOMES:
comparison of the age of our population to those of the CLEOPATRA cohort | at the inclusion
  % of patients with an age <65 years and > 65 years and <75 years and > 75 years in our study are compared to those of Cleopatra cohort
comparison of the % of patients who had a previous chemotherapy in our population to those of the CLEOPATRA cohort | at the inclusion
  % of patients with adjuvant or neo-adjuvant chemotherapy in our study are compared to those of Cleopatra cohort
comparison of the % of patients who had visceral metastasis in our population to those of the CLEOPATRA cohort | at the inclusion
  % of patients with visceral metastasis in our study are compared to those of Cleopatra cohort
comparison of the % of patients who had brain metastasis in our population to those of the CLEOPATRA cohort | at the inclusion
  % of patients with brain metastasis in our study are compared to those of Cleopatra cohort
comparison of the % of patients who had positive hormonal receptors in our population to those of the CLEOPATRA cohort | at the inclusion
  % of patients with positive hormonal receptors in our study are compared to those of Cleopatra cohort
comparison of the % of patients who had amplication of HER 2 detected in immunohistochemistry in our population to those of the CLEOPATRA cohort | at the inclusion
  % of patients with an amplication of HER 2 detected in immunohistochemistry in our study are compared to those of Cleopatra cohort
comparison of the % of patients who had a performance status >1 in our population to those of the CLEOPATRA cohort | at the inclusion
  % of patients with a performance status >1 in our study are compared to those of Cleopatra cohort
safety of the treatment: % of patient with an adverse event under treatment with grade >2 according to CTCAE | through study completion, an average of 1 year
  % of patient with an adverse event under treatment with grade >2 according to CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France